CLINICAL TRIAL: NCT04511689
Title: Comparative Study of Gene-activated Bone Substitute Based on Octacalcium Phosphate and Plasmid DNA Encoding VEGFA Gene and Xenogenic Bone Matrix for Alveolar Ridge Augmentation: an Open-label Randomized Controlled Trial
Brief Title: Comparative Study of Gene-activated Bone Substitute and Xenogenic Bone Matrix in Alveolar Ridge Augmentation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Histograft Co., Ltd. (Industry)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Other Study IDs: RU-GAM-20-05-2020
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Alveolar Bone Loss; Alveolar Ridge Pathology | Gingiva | Dental
Keywords: alveolar ridge atrophy; bone grafting; gene-activated matrix; dental implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: bone grafting with gene-activated bone substitute based on octacalcium phosphate and plasmid DNA encoding VEGFA gene mixed with autobone
  Interventions: Device: gene-activated bone substitute mixed with autobone
- control group: bone grafting with xenogenic deproteinized bone matrix mixed with autobone

INTERVENTIONS:
Device: gene-activated bone substitute mixed with autobone — gene-activated bone substitute based on octacalcium phosphate and plasmid DNA encoding VEGFA gene mixed with autobone
  Other Names: xenogenic deproteinized bone matrix mixed with autobone
  Groups: test group

SUMMARY:
The study aim is to compare the effectiveness of two bone substitutes, the gene-activated bone substitute based on octacalcium phosphate and plasmid DNA encoding VEGFA gene and xemogenic deproteinized bone matrix, mixed with shredded autobone in vertical and horizontal augmentation of alveolar ridge before dental implantation

DETAILED DESCRIPTION:
An open-label randomized controlled clinical trial, two cohort. Patients who met the inclusion criteria is planned to be enrolled into the trial. On enrollment, all patients will have screening, a set of clinical examination, instrumental investigations and laboratory tests, including dental CT of the affected jaw with the assessment of alveolar ridge width and height.

All patients enrolled in the study will be subjected to guided bone regeneration surgery of the upper or lower jaw with the use of investigational bone substitutes mixed with shredded autobone harvested during the surgery. If the height of alveolar ridge needs to be augmented, the non-resorbed systems for granular material fixation will be used.

The clinical study results will be evaluated at the time points of 1, 2, 10, 30, 90, and 180 days with clinical examination, instrumental investigations and laboratory tests. A control dental CT will be carried out before dental implantation for the primary outcome measure, at 180 days after surgery. The clinical trial completion date is the day of the second surgery, a dental implant placement. During the procedure, trephine biopsy samples will be harvested from the bone grafting area addressing the secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* partial or full edentulism;
* alveolar ridge atrophy and defects preventing from dental implant placement;
* obtained voluntary informed consent for participation in the clinical study

Exclusion Criteria:

* disability or unwillingness to give a voluntary informed consent or follow requirements of the clinical trial;
* plaque index (PI) score > 15%;
* gingival sulcus bleeding index (SBI) > 10%
* decompensated chronic diseases;
* alcohol addiction;
* a history of drug addiction;
* a history of medication with drugs affecting bone tissue metabolism;
* participation in other clinical trials (or the administration of investigational products) within 3 months prior to the study;
* conditions limiting study compliance (e.g., dementia, psycho-neurological diseases, drug addiction, and alcoholism);
* pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are subjected to guided bone regeneration surgery of the upper or lower jaw for subsequent dental implants placement.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of soft tissues (fat and fibrous) with density less then 120 HU within total volume of tissues in the bone grafting area by CT scan | 6 months
  Evaluation of the total volume of tissues in the bone grafting area using manual segmentation tool and subsequent calculation of a proportion of the low-density tissues

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | 6 months
  evaluation of the Adverse Events and Serious Adverse Events frequency
post-operative pain level | 6 months
  level of local pain assessed by Numeric rating scale (1-10)
post-operative swelling level | 6 months
  post-operative swelling level assessed by Numeric rating scale
newly formed bone tissue level | 6 months
  Volume of newly formed bone tissue in the trephine biopsy samples measured as a percentage of bone tissue in total square of histological slice

CONTACTS AND LOCATIONS:
Overall Officials: Grigory Volozhin, MD, PhD, Principal Investigator — A.I. Evdokimov Moscow State University of Medicine and Dentistry
Locations (1):
- A.I. Evdokimov Moscow State University of Medicine and Dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided